CLINICAL TRIAL: NCT04098367
Title: A Prospective, Randomized, Controlled, Multi-Center Clinical Investigation of the AcrySof IQ Vivity Extended Vision IOL vs. TECNIS Symfony and AT LARA Extended Depth of Focus IOLs
Brief Title: Clinical Investigation of the AcrySof IQ Vivity Extended Vision Intraocular Lens (IOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILI875-P001
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Aphakia
Keywords: Cataracts; Extracapsular cataract extraction; IOL; Extended depth of focus; Visual disturbances; Presbyopia; Intraocular lens
MeSH Terms: conditions — Aphakia; Cataract; Presbyopia | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- VIVITY (Experimental): VIVITY IOL implanted in the eye during cataract surgery
  Interventions: Device: VIVITY; Procedure: Cataract surgery
- SYMFONY (Active Comparator): SYMFONY IOL implanted in the eye during cataract surgery
  Interventions: Device: SYMFONY; Procedure: Cataract surgery
- AT LARA (Active Comparator): AT LARA implanted in the eye during cataract surgery
  Interventions: Device: AT LARA; Procedure: Cataract surgery

INTERVENTIONS:
Device: VIVITY — Extended vision intraocular lens intended for primary implantation for the visual correction of aphakia in adult patients with less than 1.00 diopter of preoperative corneal astigmatism in whom a cataractous lens has been removed by extracapsular cataract extraction
  Other Names: AcrySof™ IQ Vivity™ Extended Vision IOL Model DFT015
  Arms: VIVITY
Device: SYMFONY — Extended range of vision intraocular lens indicated for primary implantation for the visual correction of aphakia in adult patients with less than 1.00 diopter of pre-existing corneal astigmatism in whom a cataractous lens has been removed
  Other Names: TECNIS Symfony® Extended Range of Vision IOL Model ZXR00
  Arms: SYMFONY
Device: AT LARA — Extended depth of focus intraocular lens indicated for implantation for the visual correction of aphakia in patients with and without presbyopia in whom a cataractous lens has been removed by extracapsular cataract extraction
  Other Names: AT LARA® extended depth of focus IOL Model 829MP
  Arms: AT LARA
Procedure: Cataract surgery — Cataract removal by routine small incision surgery

SUMMARY:
The purpose of this study is to compare the visual disturbance profile of an intraocular lens (IOL) using nondiffractive optics, the VIVITY IOL, to two diffractive IOLs in subjects requiring bilateral cataract surgery. IOLs are implantable medical devices intended for long-term use over the lifetime of the cataract patient.

DETAILED DESCRIPTION:
A total of 10 scheduled visits are planned. The visits include a screening visit, 2 operative visits, and 7 postoperative visits. Both eyes will be implanted. The second eye implant will occur within 7-21 days of the first eye implant. The primary endpoint data will be collected at the Month 3 visit. Individual subject participation is expected to last 6-7 months. This study will be conducted in Australia and New Zealand.

ELIGIBILITY:
Inclusion Criteria:

* Planned cataract removal in both eyes.
* Willing and able to complete all required postoperative visits.
* Able to understand, read and write English and willing to sign an approved statement of informed consent.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential, pregnant, intend to become pregnant, breastfeeding.
* Any eye condition, disease or pathology, other than cataract, that is expected to reduce postoperative best corrected distance visual acuity, as specified in the protocol.
* Ocular trauma or ocular surface disease that would affect study measurements.
* Patients who desire monovision correction.
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Surgical, Study Director — Alcon Research, LLC
Locations (12):
- Australia (9):
  - Alcon Investigator 8047, Charlestown, New South Wales
  - Alcon Investigator 6667, Sydney, New South Wales
  - Alcon Investigator 7678, Sydney, New South Wales
  - Alcon Investigator 8052, Eastwood, South Australia
  - Alcon Investigator 7130, Hobart, Tasmania
  - Alcon Investigator 8010, Essendon, Victoria
  - Alcon Investigator 7813, Footscray, Victoria
  - Alcon Investigator 1702, Mornington, Victoria
  - Alcon Investigator 8051, Murdoch, Western Australia
- New Zealand (3):
  - Alcon Investigator 8056, Auckland
  - Alcon Investigator 8050, Auckland
  - Alcon Investigator 3656, Wellington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from nine investigative sites located in Australia and three investigative sites located in New Zealand.
Pre-assignment Details: Of the 222 enrolled, 24 subjects were exited as screen failures prior to randomization. Of the 198 subjects randomized, both eyes from five subjects and second eyes from 2 subjects (i.e., 5 first eyes, 7 second eyes) were discontinued after randomization and prior to attempted implantation. This reporting group includes all randomized and implanted subjects (193).
Period: Overall Study
Arm/Group | VIVITY | SYMFONY | AT LARA
Started | 63 | 65 | 65
First Eye Implanted | 63 | 65 | 65
Second Eye Implanted | 63 | 65 | 63
Completed | 61 | 60 | 61
Not Completed | 2 | 5 | 4
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Sick . Could not attend visit | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Implanted Analysis Set (AAS): All eyes with successful study IOL implantation in one or more eye.
Groups:
- Total: Total of all reporting groups
Arm/Group | VIVITY | SYMFONY | AT LARA | Total
Number analyzed (Participants) | 63 | 65 | 65 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (8.07) | 67.0 (9.25) | 66.1 (8.60) | 66.7 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 36 | 40 | 114
  Male | 25 | 29 | 25 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (Caucasian) | 58 | 47 | 54 | 159
  Black | 1 | 2 | 0 | 3
  Indigenous or Other Pacific Islander | 0 | 2 | 1 | 3
  Asian | 2 | 6 | 7 | 15
  Other | 2 | 8 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Not Bothered at All by Halos (QUVID Question 2.3)
Description: QUVID is a patient-reported outcomes questionnaire that collects responses from the subject about vision-related experiences. A halo is a circular spreading of light around a light source, such as car headlights at night. Question 2 of QUVID asked the subject, "In the past 7 days, have you experienced halos?" Subjects responding "No" were automatically imputed as reporting, "0=Not bothered at all." Subjects responding "Yes" were then asked Question 2.3: "In the past 7 days, how much have your halos bothered you?" Subjects responded on a 5-point scale: 0=Not bothered at all; 1=Bothered a little bit; 2=Bothered somewhat; 3=Bothered quite a bit; 4=Bothered very much. Percentage was calculated as number of subjects with score of 0 divided by number of subjects with data regardless of response, times 100.
Time Frame: Month 3 postoperative (Day 120-180 from second eye surgery)
Population: AAS with data at Month 3 postoperative visit
Measure: Number; unit: percentage of subjects
Arm/Group | VIVITY | SYMFONY | AT LARA
Number analyzed (Participants) | 63 | 65 | 63
percentage of subjects | 88.7 | 58.1 | 58.6
Statistical Analysis 1: Comparison: VIVITY vs SYMFONY; Test type: Superiority — Superiority is concluded if the lower limit of the two-sided 97.5% confidence interval exceeds zero; Miettinen-Nurminen; Difference in percentage = 30.6, 97.5% CI 2-sided [13.34 to 46.79] — VIVITY minus SYMFONY
Statistical Analysis 2: Comparison: VIVITY vs AT LARA; Test type: Superiority — Superiority is concluded if the lower limit of the two-sided 97.5% confidence interval exceeds zero; Miettinen-Nurminen; Difference in percentage = 30.1, 97.5% CI 2-sided [12.54 to 46.68] — VIVITY minus AT LARA

2. Secondary Outcome: Percentage of Subjects Not Bothered at All by Glare (QUVID Question 3.3)
Description: Glare is a wide dispersion of light, such as an intensified reflection of the sun off a glass building. Question 3 of QUVID asked the subject, "In the past 7 days, have you experienced glare?" Subjects responding "No" were automatically imputed as reporting, "0=Not bothered at all." Subjects responding "Yes" were then asked Question 3.3: "In the past 7 days, how much has your glare bothered you?" Subjects responded on a 5-point scale: 0=Not bothered at all; 1=Bothered a little bit; 2=Bothered somewhat; 3=Bothered quite a bit; 4=Bothered very much. Percentage was calculated as number of subjects with score of 0 divided by number of subjects with data regardless of response, times 100.
Time Frame: Month 3 postoperative (Day 120-180 from second eye surgery)
Population: AAS with data at Month 3 postoperative visit
Measure: Number; unit: percentage of subjects
Arm/Group | VIVITY | SYMFONY | AT LARA
Number analyzed (Participants) | 62 | 63 | 60
percentage of subjects | 53.2 | 55.6 | 35.0
Statistical Analysis 1: Comparison: VIVITY vs SYMFONY; Test type: Superiority — Superiority is concluded if the lower limit of the two-sided 97.5% confidence interval exceeds zero; Miettinen-Nurminen; Difference in percentage = -2.3, 97.5% CI 2-sided [-21.91 to 17.42] — VIVITY minus SYMFONY
Statistical Analysis 2: Comparison: VIVITY vs AT LARA; Test type: Superiority — Superiority is concluded if the lower limit of the two-sided 97.5% confidence interval exceeds zero; Miettinen-Nurminen; Difference in percentage = 8.2, 97.5% CI 2-sided [-12.00 to 27.80] — VIVITY minus AT LARA

3. Secondary Outcome: Percentage of Subjects Not Bothered at All by Starbursts (QUVID Question 1.3)
Description: A starburst is a star-shaped spreading of light around a light source, such as car headlights at night. Question 1 of QUVID asked the subject, "In the past 7 days, have you experienced starbursts?" Subjects responding "No" were automatically imputed as reporting, "0=Not bothered at all." Subjects responding "Yes" were then asked Question 1.3: "In the past 7 days, how much have your starbursts bothered you?" Subjects responded on a 5-point scale: 0=Not bothered at all; 1=Bothered a little bit; 2=Bothered somewhat; 3=Bothered quite a bit; 4=Bothered very much. Percentage was calculated as number of subjects with score of 0 divided by number of subjects with data regardless of response, times 100.
Time Frame: Month 3 postoperative (Day 120-180 from second eye surgery)
Population: AAS with data at Month 3 postoperative visit
Measure: Number; unit: percentage of subjects
Arm/Group | VIVITY | SYMFONY | AT LARA
Number analyzed (Participants) | 62 | 63 | 60
percentage of subjects | 79.0 | 55.6 | 38.3
Statistical Analysis 1: Comparison: VIVITY vs SYMFONY; Test type: Superiority — Superiority is concluded if the lower limit of the two-sided 97.5% confidence interval exceeds zero; Miettinen-Nurminen; Difference in percentage = 23.5, 97.5% CI 2-sided [4.66 to 40.86] — VIVITY minus SYMFONY
Statistical Analysis 2: Comparison: VIVITY vs AT LARA; Test type: Superiority — Superiority is concluded if the lower limit of the two-sided 97.5% confidence interval exceeds zero; Miettinen-Nurminen; Difference in percentage = 40.7, 97.5% CI 2-sided [21.16 to 57.22] — VIVITY minus AT LARA

ADVERSE EVENTS:
Time Frame: Pre-operation (Day -28) up to Day 120-180 (post second eye implantation), 6-7 months.
Description: An AE was defined at any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the test article. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. At Risk" population of preoperative and systemic AEs is reported in units of subjects; all other AE populations are reported in units of eyes.
Groups:
- Pretreatment: All subjects prior to with attempted implantation with any IOL (successful or aborted implant)
- VIVITY First Eye; VIVITY Second Eye: All eyes that had contact with the VIVITY IOL (successful or aborted implant)
- VIVITY Systemic: All subjects that had contact with the VIVITY IOL (successful or aborted implant)
- SYMFONY First Eye; SYMFONY Second Eye: All eyes that had contact with the SYMFONY IOL (successful or aborted implant)
- SYMFONY Systemic: All subjects that had contact with the SYMFONY IOL (successful or aborted implant)
- AT LARA First Eye; AT LARA Second Eye: All eyes that had contact with the AT LARA IOL (successful or aborted implant)
- AT LARA Systemic: All subjects that had contact with the AT LARA IOL (successful or aborted implant)
Arm/Group | Pretreatment | VIVITY First Eye | VIVITY Second Eye | VIVITY Systemic | SYMFONY First Eye | SYMFONY Second Eye | SYMFONY Systemic | AT LARA First Eye | AT LARA Second Eye | AT LARA Systemic
All-Cause Mortality (participants affected / at risk) | 0/193 | 0/63 | 0/63 | 0/63 | 0/65 | 0/65 | 0/65 | 0/65 | 0/63 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/193 | 1/63 | 0/63 | 0/63 | 1/65 | 3/65 | 1/65 | 3/65 | 2/63 | 4/65
Other Adverse Events (participants affected / at risk) | 0/193 | 7/63 | 7/63 | 0/63 | 12/65 | 10/65 | 0/65 | 17/65 | 16/63 | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=193) | VIVITY First Eye (N=63) | VIVITY Second Eye (N=63) | VIVITY Systemic (N=63) | SYMFONY First Eye (N=65) | SYMFONY Second Eye (N=65) | SYMFONY Systemic (N=65) | AT LARA First Eye (N=65) | AT LARA Second Eye (N=63) | AT LARA Systemic (N=65)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystoid macular oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Halo vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Posterior capsule rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paracentesis (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lens extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parathyroidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitrectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=193) | VIVITY First Eye (N=63) | VIVITY Second Eye (N=63) | VIVITY Systemic (N=63) | SYMFONY First Eye (N=65) | SYMFONY Second Eye (N=65) | SYMFONY Systemic (N=65) | AT LARA First Eye (N=65) | AT LARA Second Eye (N=63) | AT LARA Systemic (N=65)
Posterior capsule opacification (Eye disorders) | 0 (0) | 7 (7) | 7 (7) | 0 (0) | 12 (12) | 10 (10) | 0 (0) | 17 (19) | 16 (17) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT04098367/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT04098367/SAP_001.pdf